CLINICAL TRIAL: NCT02914847
Title: Imaginator: a Pilot of a Brief Functional Imagery Training Intervention for Self-harm in Young People, Supported by a Smart-phone 'App'
Brief Title: Imaginator: a Pilot of Brief Functional Imagery Training for Self-harm
Acronym: Imaginator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Martina DiSimplicio, Dr, Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/LO/1311
Record Dates: First submitted 2016-09-13; First posted 2016-09-26 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Self-Injurious Behavior
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Functional Imagery Training (FIT) (Experimental): Participants in this arm receive Functional Imagery training (FIT) immediately.
  Interventions: Behavioral: Functional Imagery Training (FIT)
- Delayed Functional Imagery Training (FIT) (No Intervention): Participants in this arm receive Functional Imagery Training (FIT) after a 3 month delay.

INTERVENTIONS:
Behavioral: Functional Imagery Training (FIT) — Functional Imagery Training comprises of three elements: a) formulation of idiosyncratic drivers of self-harming behaviour and reasons for change; b) motivational interviewing combined with mental imagery techniques that enhance motivation to change the self-harm dysfunctional habit; c) formulation of goals for change (i.e. the goal is a desired behaviour alternative to self-harm) and practice of functional imagery to support goal achievement.
  Arms: Immediate Functional Imagery Training (FIT)

SUMMARY:
Self-harm has substantial personal impacts as well as costs on the National Health Service (NHS). Around 13-17% of young people report experiences of self-harm. In Cambridgeshire, this is a significant issue with the number of admissions to hospital for self-harm in young people being higher than the United Kingdom (UK) average. Treating underlying mental illness can lead to a reduction in self-harm, but these are long interventions for complex disorders and many people who self-harm are not under treatment for mental illness. Moreover, young people struggle to access traditional mental health services where these therapies are delivered. No short interventions specifically tailored for young people have been developed so far.

The Imaginator project aims to address the urgent need for an effective and innovative short-term therapy for self-harm in young people. The investigators will pilot a new imagery-based psychological intervention for young people aged 16-25 who experience repetitive self-harm. Mental imagery (the experience of "seeing through the mind's eye") can carry intense emotions (positive and negative), and imagining something can facilitate behaviour. Imagery-based therapies have proven useful (i) for problems that feature intense, hard to manage emotions such as those associated with self-harm, and (ii) for promoting healthy behaviour. Our new intervention called Functional Imagery Training will support young people to imagine more adaptive behaviours to cope with the emotional distress that triggers self-harm, and motivate them to reduce self-harm. Imaginator will comprise of just two sessions followed by phone support over three months.

Moreover, the investigators will address the challenge of young people accessing and staying in therapy by using a smartphone app to support the therapy, as apps are widely used and favoured by this age group. The app will enable participants to continue with the strategies they have learnt in therapy by themselves, thus ensuring a potential longer-term benefit and self-empowerment.

DETAILED DESCRIPTION:
The problem of self-harm and the need short interventions for young people.

Self-harm, an "act of self-poisoning or self-injury, irrespective of the apparent purpose of the act" is a behaviour used to cope with intense emotions and psychological distress. It can occur in a variety of mental health diagnoses as well as individuals with no diagnosis. Of concern is that almost one in five young adults report self-harm behaviour. A United Kingdom (UK) survey in schools described 13% 15-16 years old had self-harmed during their life and 8% in the last year. Factors associated with self-harm include a disadvantaged socio-economic background, social isolation and lack of support, negative life events including childhood emotional, physical or sexual abuse. Although self-harm is different from suicidality, people who self-harm carry a fourfold risk of suicidal thoughts and behaviours within one year, a risk over and above risk conferred by mental health problems and psychosocial risk factors.

Self-harm has substantial personal impacts and costs on the National Health Service (NHS). In Cambridgeshire, the number of hospital admissions for self-harm has been higher than the UK average, making addressing self-harm a significant issue for local primary and secondary health care National Institute for Clinical Excellence (NICE) guidelines recommend offering a "psychological intervention that is specifically structured for people who self-harm, with the aim of reducing self-harm. In addition: (i) the intervention should be tailored to individual need, and could include cognitive-behavioural, psychodynamic or problem-solving elements; (ii) therapists should be trained and supervised in the therapy they are offering to people who self-harm; (iii) therapists should also be able to work collaboratively with the person to identify the problems causing distress or leading to self-harm." A number of interventions have been developed and have shown some efficacy at reducing self-harm in adolescents and adults. However these therapies vary between 4 sessions and much longer duration, and currently are mostly available only to individuals under mental health care after variable periods of waiting time. Moreover, almost half of young people referred recommended treatment will not attend any follow-up sessions. There is a lack of short interventions for self-harm specifically targeted at young people. Short interventions that engage young people are urgently needed to allow young people to better manage and reduce self-harm also outside secondary mental health care, and alongside / while waiting for more longterm problems to be addressed (psychiatric disorders, housing and employment difficulties etc.).

Developing new treatments for self-harm using imagery-based interventions.

Mental imagery is the process of 'seeing through the mind's eye'. Intrusive mental images carrying intense negative emotions are central to several mental disorders. For example, individuals with social anxiety will experience intrusive images of them sweating and blushing intensely while they try to speak to someone, these images will fuel their anxiety about being judged by others and possibly stop them from attending further social situations. Mental imagery associated with self-harm also appears to be a common phenomenon and individuals describe that images associated with self-harm can carry many different emotional meanings (e.g. evoking a sense of relief, or increasing the urge to self-harm), in line with what drives self-harm in every individual. The characteristics of mental images are related to the intensity of emotions and this applies to positive emotions too. For example, more vivid positive imagery has been related to greater excitement during positive mood.

Overall, this suggests that mental imagery is a common phenomenon, which many individuals are likely to experience in the context of high emotions, and that mental images could be used to generate helpful emotions. In fact, addressing distressing mental images and promoting positive imagery has been used for trauma, depression and self-harm in personality disorders. The investigators have successfully treated cases with self-harm behaviour using a short course of imagery-focused therapy for Bipolar Disorder.

Moreover, mental images can promote behaviour. Imagining something makes it more likely to act, because it simulating the actual event in the mind and it allows individuals to ''pre-experience'' all aspects the event. Hence, via imagining future scenarios individuals may feel more ready to engage in the action successfully. For example, in sports adding mental imagery training (visualising an exercise) to physical practice of an exercise improves performance. Moreover, imagining an action also involves anticipating how emotionally rewarding it is likely to be. This may enhance motivation to act. The more vivid and real-like the mental image of completing a desired action is, the stronger the positive emotion and motivation to actually do it. This type of imagery of healthy behaviour and desired actions has been developed into a therapy called Functional Imagery Training (FIT). FIT encourages individuals to imagine the benefits of working towards their goals, especially the benefits that are expected to happen right away (e.g. feeling good about oneself).

So far, FIT has been shown to be a successful approach for interventions to reduce snacking and in addictive behaviours.

Based on this, the investigators propose that FIT can train individuals to imagine more helpful behaviours rather than self-harm when distressed. FIT will train vivid and real-like imagery of alternative goals to self-harm, which is likely to produce rewarding and positive emotions. Our FIT protocol will aim to support individuals who self-harm at:

(i) identifying helpful behaviours as an alternative goal when they feel like self-harming (e.g. going for a run, listening to music); (ii) by practising mental imagery of the alternative behaviour, boosting the desire to achieve this goal; (iii) succeeding in engaging in alternative behaviours to self-harm.

Importantly, FIT will consist of two face-to-face sessions plus five brief telephone support sessions. Therefore it has the potential of offering immediate support for all those young people who are either excluded from or waiting for more complex interventions.

The challenge of engaging young people.

Imagery-based interventions focus on visual techniques and are easily amenable to be supported by a smartphone app. Smartphone usage by young people is high. Therefore, enhancing a psychological intervention via a smartphone app could be a successful strategy to ensure that young people keep practising the therapy techniques and engaging with what was learned in therapy once the sessions are over and without the need of face to face follow-up. The support of a smartphone app following the FIT sessions can aid overcome barriers to engagement reported in young people.

Therefore, the Imaginator study will tailor FIT to young people by adding a smartphone app support, which can make the intervention more interesting and approachable to this age group. The investigators have developed a bespoke app called Imaginator. This app was created collectively via six meetings of a Young People Advisory Group (YPAG: 4 members, 1 male, aged 19 to 22 years old, with a lived experience of self-harm), together with the research team and John Harper, from App Shine Development company.

In summary, self-harm behaviour is a highly prevalent problem among young people in the UK (and worldwide), and of particular urgency in Cambridgeshire. It represents a major social and healthcare problem for the community. Currently, there is a lack of short and easily accessible interventions to specifically help young people reduce self-harming behaviour. As mental imagery-based techniques have been used to reduce unwanted emotions and support motivation and helpful behaviour, The investigators propose that Functional Imagery Training (FIT) could represent a successful strategy to reduce self-harm behaviour. FIT is intended as a brief and focused intervention for young people aged 16-25 (regardless of any diagnosis) that can be added to any other pharmacological or psychological therapy. To improve access to and engagement with the intervention by young people, the investigators will deliver FIT supported by a smartphone app developed together with a Young People Advisory Group.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 - 25 years old
* Have adequate English language ability to permit the assessment and experimental measures to be completed and use of the smartphone app
* Presented with at least 2 episodes of self-harm (defined in 2.2) over the last three months
* Willing to receive support to reduce / improve management of self-harm urges and behaviour in person, over the phone and via Android smartphone app (own or made available by researchers*)
* Willing to have letters sent/phone calls made to their General Practitioner (GP) and other relevant clinicians
* Can commit to attending 2 consecutive weekly sessions, and 5 fortnightly phone follow-up sessions, and assessments over follow up period as required by the study
* Resident within geographical areas covered by the Cambridgeshire and Peterborough NHS Foundation trust (CPFT)
* Able to give consent

Exclusion Criteria:

* Experiencing current severe psychopathology that is of impediment to completing the study requirements, e.g. active psychotic symptoms (clinicians assessment)
* Currently treated under the care of the CPFT Personality Disorders Pathway
* Currently under the care of the CPFT Crisis Resolution and Home Treatment Team or under inpatient care
* Learning difficulties, organic brain disease, severe neurological impairment
* Current severe substance or alcohol abuse (clinicians assessment)
* Presence of active suicidal risk on the Mini International Neuropsychiatric Interview (MINI) confirmed by convergent clinical opinion (see risk assessment protocol, Appendix 1)
* Unwilling to engage actively in the Functional Imagery Training (FIT) intervention or to use an imagery-focused approach for treatment
* Unwilling to use a smartphone app
* Taking part in concurrent treatment studies investigating pharmacological or psychological treatment for self-harm

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Reduced Self-harm | 3 months
  Change in the presence of and number of self-reported self-harm episodes over 3 months prior to the FIT intervention to over 3 months after randomization to the FIT intervention in the Immediate FIT + Standard Care (SC) group compared to the Delayed FIT + SC group.

SECONDARY OUTCOMES:
Reduction of self-harm severity | 3 months
  Average scores on severity of self-harm ratings over 3 months
VAS reduction | 3 months
  Average scores on a Visual Analogue Scale (VAS) scale of self-efficacy ratings referred to self-harm
Imagery | 3 months
  Average scores on characteristics of mental imagery associated with self-harm when present (e.g. vividness, compellingness)
Clinical outcomes | 3 months
  Average scores on clincial questionnaire 3 months after intervention
6 month outcome self-efficacy | 6 months
  Change from pre-randomization to 6 months after intervention in average scores on self-efficacy ratings on VAS scale referring to distress associated with self-harm
Imaginator app | 3-6 months
  Correlations between endpoints scores and the following measures of Imaginator app use: number of app sessions/logins and total duration of app use, number activity cycles completed, number of personalised media uploaded, number of completed guided imagery sessions and total duration of guided imagery completed, at 3 and 6 months after the intervention.
Feasibility Data Total | 3 months
  Total number of participants referred to IMAGINATOR from different recruitment sources
Reduction of self-harm modalities | 3 months
  Average scores on self-harm modalities
Reduction of Emergency Departments (ED) visits | 3 months
  Number of Emergency Department (ED) visits
Average scores on functional outcomes | 3 months
  Average score on functional outcome
Average score on process outcome | 3 months
  Average score on process outcome measure
6 month (Emergency Department) ED visit | 6 months
  Change from pre randomisation to 6 months after intervention on number of ED attendance episodes
6 month Clinical outcome | 6 months
  Average scores on clincial questionnaire 6 months after intervention
6 month functional outcome | 6 month
  Average scores on functional outcome 6 months after intervention
6 month process outcome | 6 month
  Average scores on functional outcome 6 months after intervention
Feasibility Data Monthly | 3 month
  Monthly Recruitment Rate
Feasibility data Attrition rate | 3 month
  Attrition rate (percentage of participants completing intervention) comparing Delayed Functional Imagery Training (FIT) to Immediate FIT
Feasibility Completion | 3 month
  Completion rate of follow up assessments comparing Delayed Functional Imagery Training (FIT) to Immediate FIT

CONTACTS AND LOCATIONS:
Locations (1):
- MRC CBU, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- See also: Self-harm in over 8s guidelines — http://www.nice.org.uk/guidance/cg133
- See also: Post Traumatic Stress Disorder Management — http://www.nice.org.uk/CG26